CLINICAL TRIAL: NCT04901013
Title: A Prospective, Multicenter, Randomized, Controlled Clinical Study Of Affinity Versus SOC In The Management Of VLUs
Brief Title: Clinical Study Of Affinity Versus SOC In The Management Of VLUs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Organogenesis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-VLU-003-AFF
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Venous Leg Ulcer
Keywords: VLU; Chronic Venous Leg Ulcer; Non-healing VLU
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Affinity plus SOC (Active Comparator): Affinity is an aseptically processed, hypothermically stored fresh allograft with viable cells, growth factors/cytokines, and extracellular matrix (ECM). Affinity is human allograft tissue that is regulated as a Human Cells, Tissues, and Cellular and Tissue-Based Product (HCT/P) as defined by FDA 21 CFR Part 1271. Affinity may be applied as a wound covering to partial- and full-thickness acute and chronic wounds
  Interventions: Other: Affinity
- Standard of Care (SOC) (No Intervention): Standard of Care (SOC) includes, but is not limited to, surgical debridement, aggressive infection management, offloading, and maintenance of appropriate cleansing at the time of each dressing change.

INTERVENTIONS:
Other: Affinity — Affinity is an aseptically processed, hypothermically stored fresh allograft with viable cells, growth factors/cytokines, and extracellular matrix (ECM).
  Arms: Affinity plus SOC

SUMMARY:
This prospective, multi-center, randomized, controlled clinical study compares Affinity® plus SOC to SOC alone in subjects with VLUs. Affinity® will be used along with standard of care on venous leg ulcers (VLUs) of greater than 4 weeks which have not adequately responded to conventional ulcer therapy.

DETAILED DESCRIPTION:
Two hundred (200) subjects with a chronic VLU ranging in size from 2cm2 and 80 cm2 will be randomized 1:1 to either Affinity® and SOC or SOC alone following the 28 day screening period. Following screening and randomization, subjects shall be seen weekly for up to 24 weeks. For subjects that heal prior to week 24, a healing confirmation visit shall occur two weeks later to confirm maintenance of complete wound closure.

Subjects that are randomized into the SOC group whose VLU has not healed by week 12 may be crossed over to receive Affinity® and followed for an additional 12-14 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Ulcers of venous origin, as clinically determined by clinical signs and symptoms (e.g. hyperpigmentation of the surrounding skin, history of swelling, varicosities, lipodermatosclerosis and/or dermatitis) or other assessments (e.g. venous reflux test).
2. Venous insufficiency ulcers, of at least 1-month duration, which have not adequately responded to conventional ulcer therapy
3. Venous insufficiency ulcers between 2 cm2 and 80 cm2
4. Partial- or full-thickness VLU, including ulcers with tissue damage that extends through the epidermis and into the upper epidermis (papillary dermis), or into the deep dermis (reticular dermis) but not through muscle, tendon, capsule, or into bone.
5. Subjects are between 18 and 85 years of age.
6. IRB approved Informed Consent Form is signed before screening and treatment.
7. Subject is expected to be available for 24 week follow-up
8. Females of child-bearing potential must be practicing an acceptable means of birth control as determined by the investigator.
9. Subjects with bilateral ulcers may be enrolled.

Exclusion Criteria:

1. Ankle Brachial Index (ABI) of <0.65
2. Venous insufficiency ulcers less than 2cm2 or greater than 80cm2
3. Vasculitis, severe rheumatoid arthritis, and other collagen vascular diseases
4. Clinically significant medical conditions which would impair wound healing, as determined by the investigator, including renal, hepatic, hematologic, neurologic or immune disease
5. Signs and symptoms of infection, cellulitis, osteomyelitis
6. Necrotic or avascular ulcer beds
7. Ulcer with exposed bone, tendon or fascia
8. Subjects receiving hemodialysis or have uncontrolled diabetes
9. Subjects who are currently receiving or have received at any time within one month prior to entry into the study, corticosteroids (>15 mg/day), immunosuppressive agents, radiation therapy, or chemotherapy. Anticipated use of the above agents will exclude subjects from entry into the study.
10. Subjects enrolled in other wound drug investigational studies within the past three months, or device studies within the past 30 days.
11. Subject is pregnant or breast feeding.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-06-14 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Length of time that a wound achieves complete wound closure (CWC) | 24 weeks
  Duration (number of days) to achieve CWC from baseline to week 24 assessed between both groups

SECONDARY OUTCOMES:
Length of time that a wound achieves complete wound closure (CWC) | 12 weeks
  Duration (number of days) to achieve CWC from baseline to week 12 assessed between both groups
Greater than 40% wound closure at week 4 from baseline | 4 weeks
  Proportion of subjects achieving ≥ 40% wound closure at Week 4 from baseline
VLU improvement by or on End of Study (EOS) from baseline | 24 weeks
  Defined by >60% reduction in area, or >60% reduction in depth, or >75% reduction in volume
Incidence of ulcer recurrence | 24 weeks
  Number of recurrent ulcers
Mean number of ulcer free days | 24 weeks
  Average number of ulcer free days

CONTACTS AND LOCATIONS:
Overall Officials: Christine McLennan, Study Director — Organogenesis Inc.
Locations (1):
- ILD Research, Carlsbad, California, United States

IPD SHARING:
Plan to Share IPD: No